CLINICAL TRIAL: NCT06140836
Title: Randomized, Open-label, Multicenter, Phase 3 Trial of Repotrectinib Versus Crizotinib in Participants With Locally Advanced or Metastatic Tyrosine Kinase Inhibitor (TKI)-naïve ROS1-positive Non-Small Cell Lung Cancer (NSCLC) (TRIDENT-3)
Brief Title: A Study of Repotrectinib Versus Crizotinib in Participants With Locally Advanced or Metastatic Tyrosine Kinase Inhibitor (TKI)-naïve ROS1-positive Non-Small Cell Lung Cancer (NSCLC) (TRIDENT-3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1030; U1111-1292-0487 (Registry Identifier: WHO)
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: TKI-naïve; ROS1; NSCLC; ROS1-positive non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — repotrectinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Repotrectinib
- Arm B (Active Comparator)
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Repotrectinib — Specified dose on specified days
  Other Names: BMS-986472
  Arms: Arm A
Drug: Crizotinib — Specified dose on specified days
  Other Names: Xalkori
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of repotrectinib and crizotinib in participants with locally advanced or metastatic TKI-naïve ROS1-positive non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC
* Participant has a ROS1 gene rearrangement/fusion as detected by a local test.
* At least 1 measurable lesion according to RECIST v1.1, as assessed by the investigator.
* Participants must not be exposed previously with TKIs that demonstrated activities in ROS1-positive NSCLC
* Up to 1 prior line of systemic treatment for NSCLC is permitted
* ECOG Performance Status ≤ 2

Exclusion Criteria:

* Symptomatic brain metastases or symptomatic leptomeningeal involvement.
* History of previous cancer requiring therapy within the previous 2 years, except for NSCLC under study, squamous cell or basal-cell carcinoma of the skin, or any in situ carcinoma that has been completely resected.
* Known tumor targetable co-mutations or rearrangements
* Clinically significant cardiovascular disease (either active or within 6 months prior to enrollment)

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as per Blinded Independent Central Review (BICR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 41 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 41 months
Overall Response Rate (ORR) as per BICR according to RECIST v1.1 | Up to approximately 41 months
ORR as per Investigator according to RECIST v1.1 | Up to approximately 41 months
Duration of Response (DOR) as per BICR according to RECIST v1.1 | Up to approximately 41 months
DOR as per Investigator according to RECIST v1.1 | Up to approximately 41 months
Time to Response (TTR) as per BICR according to RECIST v1.1 | Up to approximately 41 months
TTR as per Investigator according to RECIST v1.1 | Up to approximately 41 months
PFS as per Investigator according to RECIST v1.1 | Up to approximately 41 months
Time to intracranial progressions as per BICR according to RECIST v1.1 | Up to approximately 41 months
Number of participants with Adverse Events (AEs), Serious AEs (SAEs), AEs leading to study intervention discontinuation, and drug-related AEs | Up to 30 days after last dose
Number of deaths | Up to 30 days after last dose
Number of participants without at least a 3-point change in the Non-Small Cell Lung Cancer-Symptom Assessment Questionnaire (NSCLC-SAQ) total score | Up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (122):
- United States (6):
  - Local Institution - 0221, Des Moines, Iowa
  - Local Institution - 0075, Boston, Massachusetts
  - Local Institution - 0201, Boston, Massachusetts
  - Local Institution - 0210, Mineola, New York
  - Local Institution - 0134, New York, New York
  - Local Institution - 0214, Tacoma, Washington
- Argentina (6):
  - Local Institution - 0092, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0091, ABB, Buenos Aires F.D.
  - Local Institution - 0106, Buenos Aires
  - Local Institution - 0207, Buenos Aires
  - Local Institution - 0093, Córdoba
- Local Institution - 0041, Vienna, Austria
- Brazil (11):
  - Local Institution - 0073, Belo Horizonte, Minas Gerais
  - Local Institution - 0033, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0034, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0029, Barretos, São Paulo
  - Local Institution - 0037, São José do Rio Preto, São Paulo
  - Local Institution - 0209, São Paulo, São Paulo
  - Local Institution - 0147, São Paulo, São Paulo
  - Local Institution - 0098, Rio de Janeiro
  - Local Institution - 0108, Rio de Janeiro
  - Local Institution - 0032, São Paulo
  - Local Institution - 0114, São Paulo
- Canada (2):
  - Local Institution - 0002, Toronto, Ontario
  - Local Institution - 0123, Trois-Rivières, Quebec
- Chile (2):
  - Local Institution - 0096, Viña del Mar, Región de Valparaíso
  - Fundacion Arturo Lopez Perez (FALP), Santiago, Santiago Metropolitan
- China (18):
  - Local Institution - 0168, Beijing, Beijing Municipality
  - Local Institution - 0185, Chongqing, Chongqing Municipality
  - Local Institution - 0169, Xiamen, Fujian
  - Local Institution - 0180, Guangzhou, Guangdong
  - Local Institution - 0194, Nanning, Guangxi
  - Local Institution - 0171, Harbin, Heilongjiang
  - Local Institution - 0166, Zhengzhou, Henan
  - Local Institution - 0181, Wuhan, Hubei
  - Local Institution - 0184, Changsha, Hunan
  - Local Institution - 0193, Nanjing, Jiangsu
  - Local Institution - 0202, Nanchang, Jiangxi
  - Local Institution - 0178, Changchun, Jilin
  - Local Institution - 0183, Xi'an, Shaanxi
  - Local Institution - 0186, Jinan, Shandong
  - Local Institution - 0164, Shanghai, Shanghai Municipality
  - Local Institution - 0179, Shanghai, Shanghai Municipality
  - Local Institution - 0177, Chengdu, Sichuan
  - Local Institution - 0175, Hangzhou, Zhejiang
- France (8):
  - Local Institution - 0059, Strasbourg, Alsace
  - Local Institution - 0055, Pessac, Aquitaine
  - Local Institution - 0109, Dijon, Côte-d'Or
  - Local Institution - 0057, Rouen, Haute-Normandie
  - Local Institution - 0058, La Tronche, Isère
  - Local Institution - 0189, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0060, Pierre-Bénite, Rhône
  - Local Institution - 0056, Paris
- Germany (9):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Klinikum Würzburg Mitte, Würzburg, Bavaria
  - Local Institution - 0074, Oldenburg, Lower Saxony
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Local Institution - 0035, Dresden
  - Asklepios Klinik Gauting GmbH, Gauting
  - Lungenfachklinik Immenhausen, Immenhausen
  - Marienhaus Klinikum Mainz, Mainz
- Greece (4):
  - Local Institution - 0154, Pátrai, Achaḯa
  - Local Institution - 0153, Athens, Attikí
  - Local Institution - 0155, Chaïdári, Attikí
  - "Theagenio" Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
- Local Institution - 0135, Budapest, Hungary
- India (8):
  - Local Institution - 0102, Ahmedabad, Gujarat
  - Local Institution - 0118, Ahmedabad, Gujarat
  - Local Institution - 0044, Gurugram, Haryana
  - Local Institution - 0082, Bengaluru, Karnataka
  - Local Institution - 0045, Pune, Maharashtra
  - Local Institution - 0049, Pune, Maharashtra
  - Local Institution - 0218, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0076, New Delhi, National Capital Territory of Delhi
- Italy (5):
  - Local Institution - 0151, Aviano, Friuli Venezia Giulia
  - Local Institution - 0152, Milan, Lombardy
  - Local Institution - 0149, Monza, Lombardy
  - Local Institution - 0150, Naples, Napoli
  - Local Institution - 0148, Rome, Roma
- Japan (12):
  - Local Institution - 0190, Nagoya, Aichi-ken
  - Local Institution - 0132, Kashiwa, Chiba
  - Local Institution - 0174, Matsuyama, Ehime
  - Local Institution - 0163, Sapporo, Hokkaido
  - Local Institution - 0173, Yokohama, Kanagawa
  - Sendai Kosei Hospital, Sendai, Miyagi
  - Tokyo Metropolitan Komagome Hospital, Bunkyo Ku, Tokyo
  - Local Institution - 0159, Yonago, Tottori
  - Local Institution - 0195, Fukuoka
  - Local Institution - 0160, Osaka
  - Local Institution - 0167, Osaka
  - Tokyo Metropolitan Police Hospital, Tokyo
- Local Institution - 0216, Amsterdam, North Holland, Netherlands
- Poland (2):
  - Local Institution - 0187, Lublin, Lublin Voivodeship
  - Local Institution - 0196, Olsztyn, Warmian-Masurian Voivodeship
- Romania (5):
  - Local Institution - 0030, Bucharest, București
  - Local Institution - 0066, Bucharest, București
  - Local Institution - 0031, Craiova, Dolj
  - Local Institution - 0122, Cluj-Napoca
  - Local Institution - 0067, Iași
- South Korea (5):
  - Local Institution - 0062, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0063, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (8):
  - Local Institution - 0141, A Coruña, A Coruña [La Coruña]
  - Local Institution - 0138, Santiago de Compostela, A Coruña [La Coruña]
  - Local Institution - 0140, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0137, Madrid, Madrid, Comunidad de
  - Local Institution - 0139, Majadahonda, Madrid, Comunidad de
  - Local Institution - 0142, Málaga
  - Local Institution - 0144, Seville
  - Local Institution - 0143, Valencia
- Kantonspital Baden, Baden, Canton of Aargau, Switzerland
- Turkey (Türkiye) (7):
  - Local Institution - 0086, Yenimahalle, Ankara
  - Local Institution - 0088, Adana
  - Local Institution - 0084, Ankara
  - Local Institution - 0087, Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Istanbul
  - Local Institution - 0083, Istanbul
  - Local Institution - 0085, Sakarya

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06140836.html